CLINICAL TRIAL: NCT02144974
Title: Reconstruction of the Pelvic Floor and the Vagina After Total Pelvic Exenteration Using the Transverse Musculocutaneous Gracilis Flap
Brief Title: Reconstruction of the Pelvic Floor After Total Pelvic Exenteration Using the TMG Flap
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9R025
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Reconstruction of the Pelvic Floor After Total Pelvic Exenteration.
Keywords: Total pelvic exenteration.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing total pelvic exenteration: Patients undergoing total pelvic exenteration for gynecological malignancies and reconstruction of the pelvic floor with a TMG flap.

SUMMARY:
Total pelvic exenteration (TPE) is a rare operation, which is the only possible curative intervention to treat central residual or recurrent tumors of the vulvar, vaginal, cervical, or uterine malignancies after initial surgery, radiation therapy and chemotherapy. Several options for pelvic floor and vaginal reconstruction have been described. The transverse musculocutaneous gracilis (TMG) flap has been introduced for breast reconstruction as a free flap. The investigators adopted the pedicled TMG flap for reconstruction after TPE.

Between November 2011 and February 2014, twelve patients underwent TPE and reconstruction with unilateral (6 patients) or bilateral (6 patients) pedicled TMG flaps. Five patients had vaginal reconstruction with bilateral TMG flaps. The investigators describe the operative procedure and the outcome of the operation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the department of Gynecology in the University hospital of Tampere, who underwent total pelvic exenteration with reconstruction of the pelvic floor.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the department of Gynecology in the University hospital of Tampere, who underwent total pelvic exenteration with reconstruction of the pelvic floor (no:12)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
wound healing | 6 months

SECONDARY OUTCOMES:
operative time | 1 day